CLINICAL TRIAL: NCT03790852
Title: A Phase 1/1b Open Label, Multi-center Exploratory Study to Investigate the Bioactivity, Ocular and Systemic Safety, Tolerability, and Pharmacokinetics Following Single and Multiple Intravitreal Administrations of KSI-301 in Subjects With Wet Age-Related Macular Degeneration (wAMD), Diabetic Macular Edema (DME) and Retinal Vein Occlusion (RVO)
Brief Title: Exploratory Study to Investigate the Bioactivity, Ocular and Systemic Safety, Tolerability, and Pharmacokinetics Following Single and Multiple Intravitreal Administrations of KSI-301 in Subjects With wAMD, DME and RVO
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: All patients past planned primary endpoint; decision by Sponsor to wind down open-label follow-up activities.
Sponsor: Kodiak Sciences Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: KSI-CL-101
Record Dates: First submitted 2018-12-27; First posted 2019-01-02 (Actual); Last update posted 2024-03-20 (Actual); Status verified 2022-11

CONDITIONS: Wet Age-related Macular Degeneration; Retinal Vein Occlusion; Diabetic Macular Edema
Keywords: DME; wAMD; RVO; KSI-301; Kodiak
MeSH Terms: conditions — Retinal Vein Occlusion

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- KSI-301 2.5 mg (Experimental): KSI-301 2.5 mg, 3 monthly initiating doses, with subsequent doses per protocol-specified retreatment criteria
  Interventions: Drug: KSI-301
- KSI-301 5 mg (Experimental): KSI-301 5 mg, 3 monthly initiating doses, with subsequent doses per protocol-specified retreatment criteria
  Interventions: Drug: KSI-301

INTERVENTIONS:
Drug: KSI-301 — Intravitreal injection

SUMMARY:
This is a Phase 1b open-label study to assess the bioactivity, ocular and systemic safety, tolerability, and pharmacokinetics of repeated injections of KSI-301 at two dose levels: 2.5 mg and 5 mg

ELIGIBILITY:
Inclusion Criteria:

Wet AMD Cohort

1. Treatment naïve wet age-related macular degeneration involving the fovea.
2. A lesion area <30 mm2 (12 disc areas) of any lesion type.
3. BCVA ETDRS letter score ≤ 78 and ≥ 23 (-20/25 to -20/320 Snellen equivalent) in the study eye.
4. Decrease in vision in the study eye determined by the investigator to be primarily the result of wAMD.

DME Cohort

1. Treatment naïve diabetic macular edema.
2. BCVA ETDRS letter score ≤ 78 and ≥ 23 (-20/25 to -20/320 Snellen equivalent) in the study eye.
3. Central subfield thickness (CST) of ≥ 300 microns on SD-OCT (Heidelberg Spectralis or equivalent).
4. Decrease in vision in the study eye determined by the investigator to be primarily the result of DME.

RVO Cohort

1. Treatment naïve retinal vein occlusion with macular edema and secondary visual impairment.
2. BCVA ETDRS letter score ≤ 78 and ≥ 23 (-20/25 to -20/320 Snellen equivalent) in the study eye.
3. Central subfield thickness (CST) of ≥ 300 microns on SD-OCT (Heidelberg Spectralis or equivalent).
4. Branch retinal vein occlusion (BRVO) and central retinal vein occlusion (CRVO) are both eligible.
5. Decrease in vision in the study eye determined by the investigator to be primarily the result of macular edema secondary to RVO.

General Inclusion Criteria

* Adults ≥ 21 years.

Exclusion Criteria:

Wet AMD Cohort:

1. Choroidal neovascularization due to causes other than age-related macular degeneration in the study eye.
2. Geographic atrophy and/or subretinal fibrosis involving the fovea of the study eye.
3. Prior intravitreal anti-VEGF therapy in the study eye.

DME Cohort:

1. Initial diagnosis of DME of more than 6 months from screening in the study eye.
2. Hard exudates in the fovea.
3. Prior intravitreal anti-VEGF therapy or steroid injection, or steroid implant (dexamethasone or triamcinolone) in the study eye.
4. Moderate or dense vitreous hemorrhage preventing clear. visualization of the macula or optic disc in the study eye.
5. Fibrovascular proliferation or tractional retinal detachment in the posterior pole in the study eye. If traction is present outside the posterior pole, it should be considered not at risk of increasing and threatening the macula with the use of anti-VEGF injections, in the investigator's judgement.

RVO Cohort:

1. Initial diagnosis of RVO of more than 4 months from screening in the study eye.
2. Active retinal or iris neovascularization in the study eye.
3. Prior intravitreal anti-VEGF therapy or steroid injection, or steroid implant (dexamethasone or triamcinolone) in the study eye.

For all phase 1b subjects:

1. Uncontrolled glaucoma (defined as intraocular pressure ≥ 25 mmHg despite treatment with antiglaucoma medication) in the study eye.
2. History of retinal detachment or treatment or surgery for retinal detachment in the study eye.
3. Any history of uveitis in either eye.
4. Significant media opacities, including visually significant cataract, in the study eye that might interfere with visual acuity assessments, optical coherence tomography, fundus photography, or with examination of the eye for assessment of safety.
5. Prior vitrectomy surgery in the study eye.
6. Active retinal disease other than the conditions under investigation.
7. Active ocular or periocular infection or inflammation in either eye.

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 121 (Actual)
Dates: Start 2018-12-26 (Actual); Primary Completion 2021-06-02 (Actual); Study Completion 2022-06-09 (Actual)

PRIMARY OUTCOMES:
Incidence of ocular (study eye) and systemic adverse events | Week 72

OTHER OUTCOMES:
Mean change in central retinal thickness on optical coherence tomography | Baseline, Week 72
Mean change in best corrected visual acuity | Baseline, Week 72

CONTACTS AND LOCATIONS:
Overall Officials: Pablo Velazquez-Martin, MD, Study Director — Kodiak Sciences Inc
Locations (11):
- United States (11):
  - Retinal Research Institute, LLC, Phoenix, Arizona
  - Retina Vitreous Associates Medical Group, Beverly Hills, California
  - Northern California Retina Vitreous Associates, Mountain View, California
  - Byers Eye Institute at Stanford, Palo Alto, California
  - Retina Vitreous Associates of Florida, St. Petersburg, Florida
  - Sierra Eye Associates, Reno, Nevada
  - Mid Atlantic Retina, Philadelphia, Pennsylvania
  - Retina Research Institute of Texas, Abilene, Texas
  - Austin Clinical Research, Austin, Texas
  - Retina Consultants of Texas, Bellaire, Texas
  - Retina Consultants of Texas Woodlands, The Woodlands, Texas